CLINICAL TRIAL: NCT04791800
Title: Evaluation of the Clinical Performance of the STANDARD™ Q Malaria/CRP Duo Test (SD Biosensor, South Korea) for the Diagnosis of Malaria and the Detection of C-reactive Protein (CRP) in Fingerprick Blood of Febrile Patients
Brief Title: Clinical Evaluation of the STANDARD™ Q Malaria/CRP Duo Test
Status: Completed | Type: Observational
Sponsor: Foundation for Innovative New Diagnostics, Switzerland (Other)
Collaborators: National Institute of Malaria Research, New Delhi, India (Unknown)
Responsible Party: Sponsor
Other Study IDs: 8820-2/1
Record Dates: First submitted 2020-08-10; First posted 2021-03-10 (Actual); Last update posted 2021-03-10 (Actual); Status verified 2021-03

CONDITIONS: Fever Malaria
Keywords: malaria; fever; C-reactive protein; point-of-care testing
MeSH Terms: conditions — Malaria; Fever

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Malaria/CRP combination test — Testing with a malaria/CRP combination test, in parallel with a standard malaria RDT (to guide case management), preparation of thin/thick films for expert malaria microscopy, and collection of venous blood for subsequent CRP quantification.

SUMMARY:
The aim of this study is to assess the clinical performance (sensitivity, specificity, positive and negative predictive values) of the STANDARD™ Q Malaria/CRP Duo Test when used by health care workers (HW) in a point of care (POC) setting in malaria endemic areas in India. Performance will be assessed in comparison with expert microscopy as the reference test for malaria, and with a high quality, commercially available C-Reactive Protein (CRP) test kit run on a laboratory machine as a reference test for CRP.

ELIGIBILITY:
Inclusion Criteria:

* clinically suspected malaria on the basis of fever or history of fever in the previous 72 h
* age ≥ 5 years, (iii) having been informed of the study and signed a written consent form

Exclusion Criteria:

* signs of severe malaria or other severe disease
* patients not fulfilling the inclusion criteria.

Min Age: 5 Years | Sex: All
Age Groups: Child, Adult, Older Adult
Study Population: Patients aged 5 years and above with clinically suspected malaria on the basis of fever or history of fever in the previous 72 h, either enrolled by passive case detection in health care facilities, or by active case detection in the surrounding communities.
Sampling Method: Non-Probability Sample
Enrollment: 1808 (Actual)
Dates: Start 2019-04-08 (Actual); Primary Completion 2020-03-16 (Actual); Study Completion 2020-09-01 (Actual)

PRIMARY OUTCOMES:
Clinical performance of the Malaria/CRP combination test for malaria diagnosis at day 0 | Day 0
  Point estimates (with 95% confidence intervals) of the sensitivity, specificity, positive and negative predictive values of the STANDARD™ Q Malaria/CRP Duo Test for the diagnosis of malaria, in comparison with expert microscopy as the reference test at day 0 (first day of presentation).
Clinical performance of the Malaria/CRP combination test for detection of high levels of C-reactive protein at day 0 | Day 0
  Point estimates (with 95% confidence intervals) of the sensitivity, specificity, positive and negative predictive values of the STANDARD™ Q Malaria/CRP Duo Test for the detection of CRP at day 0, in comparison with the CRP-LX reagent kit used with the Roche Diagnostics Cobas™ c111 chemistry analyser, or equivalent, as the reference test.

CONTACTS AND LOCATIONS:
Overall Officials: Anupkumar Anvikar, MD, Principal Investigator — National Institute of Malaria Research, New Delhi, India
Locations (1):
- NIMR, New Delhi, India

IPD SHARING:
Plan to Share IPD: No